CLINICAL TRIAL: NCT00170794
Title: A One Year, Multicenter, Open-Label, Single Arm, Pilot Study of the Renal Safety of Everolimus in Addition to Cyclosporine Microemulsion in Cardiac Transplant Recipients.
Brief Title: Renal Safety of Everolimus in Addition to Cyclosporine Microemulsion in Cardiac Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001A2412
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Cardiac Transplantation
Keywords: cardiac transplantation, everolimus, cyclosporine microemulsion, GFR
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus (RAD001)

SUMMARY:
The purpose of the study is to determine the extent of cyclosporine microemulsion dose reduction required to maintain stable renal function in maintenance cardiac transplant recipients, after initiation of everolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cardiac transplant recipients, 18-70 years old, with established cardiac allograft vasculopathy or at risk to develop a cardiac allograft vasculopathy.
* Patients who are more than 12 months post-transplant and who are receiving a cyclosporine microemulsion-based immunosuppressive regimen with/without azathioprine /mycophenolate mofetil, with/without steroids.
* Patients need to have stable renal function with a calculated GFR exceeding 40 ml/min (Nankivell).
* Patients without a biopsy-proven acute rejection ≥ grade 2, within 12 months prior to study entry.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment. Effective contraception must be used during the trial and for 4 weeks following discontinuation of the study medication, even where there has been a history of infertility.
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria:

* Patients who are recipients of multiple solid organ transplants.
* Patients with a calculated GFR of less than 40 ml/min.
* Patients with a biopsy-proven acute rejection episode ≥ 2 within 12 months prior to study entry.
* Patients who had received any investigational drug within 4 weeks prior to study entry.
* Patients currently being treated with sirolimus or having a history of prior therapy or having a hypersensitivity to drug similar to everolimus.
* Patient with a platelet count of < 50,000/mm3 or with a white blood cell count of ≤ 2,500/mm3 or with a hemoglobin value < 10 g/dL.
* Presence of severe hypercholesterolemia (≥ 9.1 mmol/L) or hypertriglyceridemia (≥ 8.55 mmol/L).
* Patient with NYHA class IV heart failure, or with left ventricular ejection fraction <30%. Patients with life-threatening cardiac allograft vasculopathy and/or graft dysfunction (life expectancy 1 year).
* Patients with severe systemic infections.
* Patients who are known to have HBsAg or HCV positive hepatitis, or who are HIV positive. Serology results obtained within 6 months prior to study entry are acceptable. If results cannot be obtained prior to study entry, a sample must be retained for later analysis. This stored sample will be destroyed at the end of study.
* Patients with any past (within the last 5 years) or present malignancy other than non-melanotic skin cancer.
* Existence of a co-morbid condition likely to result in death prior to study completion
* Symptoms of significant mental illness, which in the opinion of the investigator may interfere with the patient's ability to comply with the protocol. History of drug or alcohol abuse within 1 year of baseline.
* Inability to cooperate or communicate with the investigator.
* Female patients of childbearing potential who are planning to become pregnant, who are pregnant and/or lactating, or who are unwilling to use effective means of contraception.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Comparing calculated glomerular filtration rate (GFR) at Month 3 (Week 12) to Baseline and by comparing the daily cyclosporine dose at Month 3 (Week 12) to Baseline.

SECONDARY OUTCOMES:
Incidence of acute rejection episode greater than or equal to grade 3A.
Safety laboratory tests including lipid profiles, hematology and proteinuria.
Incidence of premature study treatment discontinuation.
Incidence of serious adverse avents (SAEs).
Incidence of admission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Result] Ross H, Pflugfelder P, Haddad H, Cantarovich M, White M, Ignaszewski A, Howlett J, Vaillancourt M, Dorent R, Burton JR; CADENCE Study Group (CAnadian Pilot Sutdy to Determine Safe and Effective Dosing of Neoral and CErtican in Stable Cardiac Transplant Recipients). Reduction of cyclosporine following the introduction of everolimus in maintenance heart transplant recipients: a pilot study. Transpl Int. 2010 Jan;23(1):31-7. doi: 10.1111/j.1432-2277.2009.00940.x. PMID 20050127